CLINICAL TRIAL: NCT02902653
Title: Efficacy and Safety of Hourly Titrated Misoprostol Versus Vaginal Dinoprostone and Misoprostol for Cervical Ripening and Labor Induction: Randomized Clinical Trial
Brief Title: Efficacy and Safety of Hourly Titrated Misoprostol Versus Vaginal Dinoprostone and Misoprostol for Cervical Ripening and Labor Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oihane Lapuente Ocamica (Other Government)
Responsible Party: Sponsor-Investigator, Oihane Lapuente Ocamica, Medical Doctor, Basque Health Service
Organization: Basque Health Service (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV-MV-MO
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Labor, Induced
Keywords: misoprostol; dinoprostonal; induction
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral misoprostol (Experimental): Administration of oral misoprostol according to a "3x1" diagram, that is,3 oral doses (1 per hour) and then 1 hour without treatment
  Interventions: Drug: Oral misoprostol
- Vaginal misoprostol (Active Comparator): vaginal misoprostol, 25 microgs every 4 hours
  Interventions: Drug: Vaginal misoprostol
- Vaginal dinoprostone (Active Comparator): vaginal dinoprostone, 10 mg during 24 hours (maximum)
  Interventions: Drug: Vaginal dinoprostone

INTERVENTIONS:
Drug: Oral misoprostol — hourly titrated misoprostol
  Arms: Oral misoprostol
Drug: Vaginal misoprostol — Administration of 25 microgs every 6 hours, maximum 150 microgr
  Arms: Vaginal misoprostol
Drug: Vaginal dinoprostone — Vaginal delivery system of 10mg of dinoprostone
  Arms: Vaginal dinoprostone

SUMMARY:
This study evaluates the efficacy and safety of the administration of oral misoprostol versus vaginal dinoprostone and vaginal misoprostol for cervical ripening and labor induction.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* single pregnancy
* cephalic presentation
* intact membranes
* unfavorable cervix ( less than 6 Bishop )
* CTGR not reactive decelerative
* Signed informed consent by the patient.

Exclusion Criteria:

* prior Cesarean section or previous uterine surgery .
* Allergy or intolerance to any of the study drugs
* stillbirth
* uterine growth restricted fetuses
* contraindication for vaginal delivery
* Anterior placenta
* Multiparity
* moderate to severe heart disease
* hypertensive disorders of pregnancy
* Suspected chorioamnionitis
* Coagulation disorders
* history of epileptic seizures
* liver or kidney disease
* Cognitive impairment or bad knowledge of Spanish

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 372 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Compare the percentage of women in each group who achieved vaginal delivery within 24 hours after the beginning of administration in each group (oral misoprostol, vaginal misoprostol and intravaginal dinoprostone) | 24 hours

SECONDARY OUTCOMES:
The number of women who manage cervical favorable conditions at 12 hours after the beginning of administration in each group | 12 hours
The number of women who manage cervical favorable conditions at 24 hours after the beginning of administration in each group | 24 hours
The percentage of women in each group who achieved vaginal delivery at 12 hours after the beginning of administration in each group | 12 hours
Compare the number of women who achieve a vaginal delivery in the 3 groups (oral misoprostol, vaginal misoprostol and intravaginal dinoprostone) | 24 hours
The number of caesarean sections in each group (oral misoprostol, vaginal misoprostol and intravaginal dinoprostone) | 24 hours
Compare the percentage of women requiring oxytocin in each group | 24 hours
The percentage of women in each group having tachysystole | 24 hours
Compare the number of women suffering from uterine rupture in each group | 24 hours
The percentage of women in each branch having uterine hypertonia | 24 hours
Maternal morbility-mortality among pregnant participants | up to 180 days
Compare fetal or neonatal morbility-mortality among the 3 groups | up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Oihane Lapuente Ocamica, Principal Investigator — OIHANE.LAPUENTEOCAMICA@osakidetza.eus
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Basque Country, Spain

REFERENCES:
- [Derived] Lapuente-Ocamica O, Ugarte L, Lopez-Picado A, Sanchez-Refoyo F, Lasa IL, Echevarria O, Alvarez-Sala J, Farinas A, Bilbao I, Barbero L, Vicarregui J, Hernanz Chaves R, Paz Corral D, Lopez-Lopez JA. Efficacy and safety of administering oral misoprostol by titration compared to vaginal misoprostol and dinoprostone for cervical ripening and induction of labour: study protocol for a randomised clinical trial. BMC Pregnancy Childbirth. 2019 Jan 8;19(1):14. doi: 10.1186/s12884-018-2132-3. PMID 30621614